CLINICAL TRIAL: NCT01584817
Title: A Repeated Instruction by Telephone on the Day Before Colonoscopy Improves the Quality of Bowel Preparation and Colonoscopy Procedure : a Prospective Randomized, Controlled Trial
Brief Title: A Repeated Instruction by Telephone on the Day Before Colonoscopy to Patients Undergoing Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 20120405-6
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Ottawa Score; Adenoma
Keywords: colonoscopy; bowel preparation; education
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal education (No Intervention): patients in this arm was educated about bowel preparation on the day of reservation by nurse for 15 minutes and meanwhile a booklet was also sent to them.
- telephone education (Other): A repeated instruction by telephone on the day before colonoscopy was conducted
  Interventions: Other: telephone education

INTERVENTIONS:
Other: telephone education — A repeated instruction by telephone on the day before colonoscopy was conducted
  Arms: telephone education

SUMMARY:
Cell phone retell the instruction of bowel preparation on the day before colonoscopy would help patient to prepare for colonoscopy and improve the quality of the bowel preparation.

DETAILED DESCRIPTION:
Colonoscopy is the gold standard in the diagnosis of colorectal disease. The success of colonoscopy depends on high-quality bowel preparation by patients. Inadequate bowel cleansing reduces the speed, the cecal intubation rate, and the number of polyps detected. It also increases costs, mostly due to repeated procedures. The quality of bowel cleansing has remained suboptimal even though numerous different products and regimens have been tested and compared in no fewer than six meta-analyses. Therefore, a completely different approach to improve precolonoscopy bowel cleansing is welcome.

There are many factors effect the bowel preparation such as age, cirrhosis diabetes, drug compliance, cerebral infarction, dementia, history of major surgery. 20% of patients with poor bowel preparation were due to bad compliance. Studies found that addressing patient perceptions with an inexpensive and simple booklet based on the Health Belief Model improved preparation quality. We assume that doctor retelling the instruction of bowel preparation by cell phone on the day before colonoscopy would help patient to prepare for colonoscopy and improve the quality of the bowel preparation.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing colonoscopy

Exclusion Criteria:

* disturbance of water and electrolyte
* history of colorectal surgery
* severe colonic stricture or obstructing tumor
* known or suspected bowel obstruction or perforation
* toxic colitis or megacolon
* dysphagia
* compromised swallowing reflex or mental status
* significant gastroparesis or gastric outlet obstruction or ileus
* severe chronic renal failure (creatinine clearance <30 mL/minute)
* severe congestive heart failure (New York Heart Association class III or IV)
* uncontrolled hypertension (average systolic blood pressure >170 mm Hg, average diastolic blood pressure >100 mm Hg)
* pregnant or lactating women
* patients who cannot give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation quality at the time of colonoscopy defined by Ottawa score<6 | up to 3 months
  Ottawa score：A)cleanliness of each part of the colon: 0=excellent 1=good 2=fair 3=poor 4=inadequate B)fluid in whole colon: small=0 moderate=1 large=2
  The bowel preparation was considered inadequate if (1) inadequate visualization on colonoscopy defined by Ottawa score≥6; (2) the colonoscopy was cancelled because of poor bowel preparation or personal reasons; (3) incomplete colonoscopy.

SECONDARY OUTCOMES:
Cecum intubation time | up to 3 months
  Total time of colonoscope intubation from anus to cecum
Withdrawal time | up to 3 months
  Total time of colonoscope intubation from cecum to anus
Polyp detection rate | up to 3 months
  The proportion of participants with at least one polyp in each group
Compliance rate to instruction | up to 3 months
  The proportion of participants compliance to instruction of bowel preparation
Willingness undergo a repeated bowel preparation | up to 3 months
  The number of patients have a willingness to undergo a repeated bowel preparation if needed

CONTACTS AND LOCATIONS:
Overall Officials: pan yanglin, MD., Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Liu X, Luo H, Zhang L, Leung FW, Liu Z, Wang X, Huang R, Hui N, Wu K, Fan D, Pan Y, Guo X. Telephone-based re-education on the day before colonoscopy improves the quality of bowel preparation and the polyp detection rate: a prospective, colonoscopist-blinded, randomised, controlled study. Gut. 2014 Jan;63(1):125-30. doi: 10.1136/gutjnl-2012-304292. Epub 2013 Mar 16. PMID 23503044